CLINICAL TRIAL: NCT07122895
Title: Sex Differences in NMDA-enhancing Treatment of Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH114-REC3-042
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; NMDA; Negative symptoms; Sex difference
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMDAE (Experimental): An NMDA enhancer
  Interventions: Drug: NMDAE
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Cap

INTERVENTIONS:
Drug: NMDAE — Use of an NMDA enhancer for the treatment of negative symptoms
  Arms: NMDAE
Drug: Placebo Cap — Use of placebo as a comparator
  Arms: Placebo

SUMMARY:
Schizophrenia differs between sexes in clinical symptoms and functional outcome. Negative symptoms are the core pathology of this disease. NMDA receptor (NMDAR) dysfunction is a key factor in negative symptoms. This study aims to examine the sex difference in the efficacy of an NMDA-enhancer (NMDAE) for the treatment of negative symptoms in schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia differs between sexes in clinical symptoms and functional outcome. Negative symptoms, the core pathology of this disease, principally determine the patients' prognoses. NMDAR dysfunction is a key factor in negative symptoms. Whether NMDAR-enhancing treatment can improve negative symptoms and whether there is sex difference need to be studied. The subjects are the schizophrenia patients with predominantly negative symptoms. They will continue their original treatment and be double-blindly, randomly assigned to receive 12-week: (1) NMDAE (N = 60), or (2) placebo (N = 30). There will be half men and half women in each group. We will measure clinical manifestations and side effects at weeks 0, 4, 8, and 12 using Scale for Assessment of Negative Symptoms (the primary outcome), Positive and Negative Syndrome Scale-negative subscale, Clinical Global Impression, Quality of Life Scale, Global Assessment of Function, and scale of side effects. At week 0 and week 12, we will assess 7 cognitive domains. Chi-square (or Fisher's exact test) will be used to compare differences of categorical variables and t-test (or Mann-Whitney test if the distribution is not normal) for continuous variables between treatment groups. Mean changes from baseline in repeated-measure assessments will be assessed using the generalized estimating equation (GEE). All p values for clinical measures will be based on two-tailed tests with a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Have a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of schizophrenia
* keep stable mentally for ≥ 6 months before baseline and meet the following clinical criteria: predominantly negative symptoms for ≥ 6 months, a minimum baseline total score of 40 on the SANS, a minimum baseline score of 24 on the negative subscale of the PANSS, and a maximum score of 3 on each item of PANSS-positive subscale;
* Are physically healthy and laboratory assessments (including blood routine, biochemical tests) are clinically insignificant;
* Have been keeping a fixed dose of antipsychotics for at least 6 months, and that is not allowed to change during the 12-week study period
* Have sufficient education to communicate effectively and are capable of completing the assessments of the study
* Agree to participate in the study and provide written informed consent

Exclusion Criteria:

* DSM-5 diagnosis of intellectual disability or substance (including alcohol) use disorder
* History of epilepsy, head trauma, or serious medical or central nervous system diseases (other than schizophrenia) which may interfere with the study
* Clinically evident depressive symptoms or a baseline score>7 on the Hamilton Depression Rating Scale-17 items
* Clinically relevant parkinsonism or a baseline score >3 on the sum of the first eight items of the Simpson-Angus Scale (SAS)
* Pregnancy or lactation
* Inability to follow protocol

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Change of scales for the Assessment of Negative Symptoms (SANS) total score | week 0, 4, 8, 12
  Assessment of negative symptoms. Minimum value: 0, maximum value:100, the higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change of Negative subscale of PANSS | week 0, 4, 8, 12
  Assessment of negative symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
Change of Clinical Global Impression | Frame: week 0, 4, 8, 12
  Assessment of general impression. Minimum value: 1, maximum value:7, the higher scores mean a worse outcome.
Change of Global Assessment of Functioning composite | week 0, 4, 8, 12
  Assessment of social, occupational, and psychological function. Minimum value: 1, maximum value:100, the higher scores mean better function.
Change of Quality of Life Scale | week 0, 4, 8, 12
  Assessment of life quality. Minimum value: 0, maximum value:126, the higher scores mean a better outcome.
Change of cognitive function composite | Week 0, 12
  Ten tests for assessment of 7 cognitive domains:
  1. speed of processing (assessed by Category Fluency, Trail Marking A, WAIS-III Digit Symbol-Coding)
  2. sustained attention (Continuous Performance Test)
  3. working memory: verbal (digit span) and nonverbal (spatial span)
  4. verbal learning and memory (WMS-III, word listing)
  5. visual learning and memory (WMS-III, visual reproduction)
  6. reasoning and problem solving (WISC-III, Maze)
  7. social cognition (MSCEIT) For the domain (a. and c.) with more than one test, a composite T score will be calculated by standardizing the average of each T score. Furthermore, a global composite score (for all seven domains) and a neurocognitive composite score (for the first 6 domains) will be also calculated by standardizing the average of the T score of each domain (Lane HY et al, JAMA Psychiatry 2013)

OTHER OUTCOMES:
Change of Positive and Negative Syndrome Scale (PANSS) | week 0, 4, 8, 12
  Assessment of overall symptoms. Minimum value: 30, maximum value:210, the higher scores mean a worse outcome.
Change of Positive subscale of PANSS | Frame: week 0, 4, 8, 12
  Assessment of positive symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
Change of General Psychopathology subscale of PANSS | week 0, 4, 8, 12
  Assessment of general psychopathology. Minimum value: 16, maximum value:112, the higher scores mean a worse outcome.
Change of Hamilton Rating Scale for Depression | week 0, 4, 8, 12
  Assessment of depressive symptoms. Minimum value: 0, maximum value:52, the higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan